CLINICAL TRIAL: NCT06989632
Title: Total Lumbar Disc Prosthesis and Subsequent Work Activity 5 Years After Total Lumbar Disc Replacement
Brief Title: Total Lumbar Disc Prosthesis and Subsequent Work Activity at at Least Five Years After Total Lumbar Disc Replacement
Status: Recruiting | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Vicente Vanaclocha, Associate Professor of Surgery, University of Valencia
Other Study IDs: 19/2024
Record Dates: First submitted 2025-01-09; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-05

CONDITIONS: Lumbar Disc Degeneration; Lumbar Disc Disease; Sciatica; Lumbar Disc Herniation; Lumbar Degenerative Disease
Keywords: Chronic low back pain; Total lumbar disc replacement; Total lumbar disc arthroplasty; Sciatica
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral disc disease; Sciatica; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Total Lumbar Disc replacement: These patients have been submitted to total lumbar disc replacement and we want to know the work and sportive activities they are able to undertake in the years after the total lumbar disc replacement
  Interventions: Device: We want to know the work and sport activities that our patients are able to undertake after a total lumbar disc replacement

INTERVENTIONS:
Device: We want to know the work and sport activities that our patients are able to undertake after a total lumbar disc replacement

SUMMARY:
Lumbosciatica is a very prevalent pathology. When conservative treatments fail, surgery should be considered. The traditional surgical treatment is lumbar arthrodesis. The vast majority of patients who undergo spinal fusion cannot return to their same job and a good number of them never work again. Another form of treatment for lumbosciatica is the implantation of a lumbar disc prosthesis. This technique preserves the mobility of the lumbar area that has been operated on. This allows for a greater return to work and a higher percentage of those who return to the same job. This study aims to quantify how many of the patients who have had a lumbar disc prosthesis implanted in the last twenty years have returned to their same job, how many have had to change their jobs, and how many have not returned to work and are now totally or completely disabled from work.

DETAILED DESCRIPTION:
Low back pain is one of the most prevalent pathologies in the world population and one of the most frequent causes of temporary and permanent work incapacity, particularly in today's largely sedentary society.

Although its etiology is broad, degenerative disc disease, herniated disc, and osteoarthritis of the facet joints are its most common causes.

Conservative treatments resolve many cases, but when they are not effective, surgical options must be considered. These can be classified into two groups: those involving vertebral fusion with loss of mobility at the level or levels in question and those attempting to preserve it.

In lumbar disc herniation, the classic treatment, discectomy, consists of more or less completely removing the nucleus pulposus through a relatively small posterior annulotomy. This causes a loss of height of the intervertebral disc and the foramina and overload of the articular facets, which over time can be accompanied by arthritic changes and trigger chronic lumbar pain.

In the degeneration of the intervertebral disc and the osteoarthritis of the articular facets, the traditional surgical technique is the arthrodesis of the vertebral segment or segments causing the symptoms. The immobilization of the painful spinal area limits the progression of the foraminal stenosis and the overload of the articular facets of the level or levels operated on. However, the fusion alters the biomechanics of the spine, causing the overload of the adjacent vertebral segments with degeneration and osteoarthritis of these, which is the cause of chronic pain. It is not uncommon that, over the years, reintervention is required to extend the arthrodesis. In turn, a larger area of fused spine will cause more overload of the adjacent levels, which will also suffer the same process of degeneration and arthrosis mentioned above, thus creating a vicious circle.

The initial step of fusion of the painful joint has also been followed in the spine in the attempt to preserve mobility by implanting a complete prosthesis of the intervertebral disc, provided that there is no degeneration or arthrosis of the articular facets. It is an option to consider compared to arthrodesis of the same segment with the appropriate surgical technique (posterolateral arthrodesis, PLIF, TLIF, X-LIF, ALIF, OLIF, 360º lumbar arthrodesis, etc.).

Studies comparing lumbar arthrodesis and arthroplasty indicate that complete lumbar disc prostheses provide a better quality of life, better control of lumbar and radicular pain symptoms, an earlier return to work, a lower incidence of adjacent level syndromes, and a lower number of complications and reinterventions. These differences are most noticeable during the first year after surgery, disappear after two years, and reappear after five years, due to the appearance of adjacent level syndrome. However, we have been able to find in the scientific literature after a thorough search which of the two surgical techniques, arthrodesis or arthroplasty at the lumbar level, achieves a greater return to the same job, or even if there are differences in terms of the work activity that each of the two surgical techniques allows. The objective of the present study is to first analyze in patients with complete lumbar disc prosthesis the percentage of return to the same job, of work activity even if it is in another job, if there is a change of work activity to what type it is changed and finally the percentage of patients who are left with work disability, of what kind and with what degree of disability. To compare with lumbar arthrodesis is not possible at this time because the arthrodesis technique, unlike arthroplasty, is very variable according to the surgeons on the team, and in our Institution, it is not possible to obtain retrospectively a homogeneous group with which to compare.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years with symptomatic lumbar degenerative disc herniation and/or lumbar disc herniation.

Exclusion Criteria:

* Any patient who BEFORE the implantation of a complete lumbar disc prosthesis had undergone any other type of surgical intervention on the lumbar spine. In particular, patients who had previously undergone a discectomy, whatever its form, or a spinal arthrodesis, whatever its technique, will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic lumbar degenerative disc herniation and/or lumbar disc herniation that underwent a total lumbar disc replacement
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2006-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have had a lumbar disc prosthesis implanted in the last twenty years and have returned to their same job | We started to implant total lumbar disc prosthesis in 2006 and have continued up to now. We want to know the results in our patients re work and sport activities at 01 May 2025
  Percentage of participants who have not returned to work and are now totally or completely disabled from work

CONTACTS AND LOCATIONS:
Locations (1):
- Consorcio Hospital General Universitario de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skold C, Tropp H, Berg S. Five-year follow-up of total disc replacement compared to fusion: a randomized controlled trial. Eur Spine J. 2013 Oct;22(10):2288-95. doi: 10.1007/s00586-013-2926-y. Epub 2013 Jul 29. PMID 23893083
- [Background] Wei J, Song Y, Sun L, Lv C. Comparison of artificial total disc replacement versus fusion for lumbar degenerative disc disease: a meta-analysis of randomized controlled trials. Int Orthop. 2013 Jul;37(7):1315-25. doi: 10.1007/s00264-013-1883-8. Epub 2013 May 4. PMID 23645003
- [Background] Berg S, Tullberg T, Branth B, Olerud C, Tropp H. Total disc replacement compared to lumbar fusion: a randomised controlled trial with 2-year follow-up. Eur Spine J. 2009 Oct;18(10):1512-9. doi: 10.1007/s00586-009-1047-0. Epub 2009 Jun 9. PMID 19506919
- [Background] Eliasberg CD, Kelly MP, Ajiboye RM, SooHoo NF. Complications and Rates of Subsequent Lumbar Surgery Following Lumbar Total Disc Arthroplasty and Lumbar Fusion. Spine (Phila Pa 1976). 2016 Jan;41(2):173-81. doi: 10.1097/BRS.0000000000001180. PMID 26751061
- [Background] Radcliff K, Spivak J, Darden B 2nd, Janssen M, Bernard T, Zigler J. Five-Year Reoperation Rates of 2-Level Lumbar Total Disk Replacement Versus Fusion: Results of a Prospective, Randomized Clinical Trial. Clin Spine Surg. 2018 Feb;31(1):37-42. doi: 10.1097/BSD.0000000000000476. PMID 28005616
- [Background] Song J, Katz A, Ngan A, Silber JS, Essig D, Qureshi SA, Virk S. Comparison of value per operative time between anterior lumbar interbody fusion and lumbar disc arthroplasty: A propensity score-matched analysis. J Craniovertebr Junction Spine. 2022 Oct-Dec;13(4):427-431. doi: 10.4103/jcvjs.jcvjs_99_22. Epub 2022 Dec 7. PMID 36777911
- [Background] Zigler J, Gornet MF, Ferko N, Cameron C, Schranck FW, Patel L. Comparison of Lumbar Total Disc Replacement With Surgical Spinal Fusion for the Treatment of Single-Level Degenerative Disc Disease: A Meta-Analysis of 5-Year Outcomes From Randomized Controlled Trials. Global Spine J. 2018 Jun;8(4):413-423. doi: 10.1177/2192568217737317. Epub 2017 Nov 16. PMID 29977727
- [Background] Ding F, Jia Z, Zhao Z, Xie L, Gao X, Ma D, Liu M. Total disc replacement versus fusion for lumbar degenerative disc disease: a systematic review of overlapping meta-analyses. Eur Spine J. 2017 Mar;26(3):806-815. doi: 10.1007/s00586-016-4714-y. Epub 2016 Jul 23. PMID 27448810
- [Background] Mattei TA, Beer J, Teles AR, Rehman AA, Aldag J, Dinh D. Clinical Outcomes of Total Disc Replacement Versus Anterior Lumbar Interbody Fusion for Surgical Treatment of Lumbar Degenerative Disc Disease. Global Spine J. 2017 Aug;7(5):452-459. doi: 10.1177/2192568217712714. Epub 2017 Jul 7. PMID 28811990
- [Background] Geisler FH. Surgical treatment for discogenic low-back pain: lumbar arthroplasty results in superior pain reduction and disability level improvement compared with lumbar fusion. SAS J. 2007 Feb 1;1(1):12-9. doi: 10.1016/SASJ-2006-0002-RR. eCollection 2007. PMID 25802574
- [Background] Mu X, Wei J, A J, Li Z, Ou Y. The short-term efficacy and safety of artificial total disc replacement for selected patients with lumbar degenerative disc disease compared with anterior lumbar interbody fusion: A systematic review and meta-analysis. PLoS One. 2018 Dec 28;13(12):e0209660. doi: 10.1371/journal.pone.0209660. eCollection 2018. PMID 30592739
- [Background] Bai DY, Liang L, Zhang BB, Zhu T, Zhang HJ, Yuan ZG, Chen YF. Total disc replacement versus fusion for lumbar degenerative diseases - a meta-analysis of randomized controlled trials. Medicine (Baltimore). 2019 Jul;98(29):e16460. doi: 10.1097/MD.0000000000016460. PMID 31335704
- [Background] Cui XD, Li HT, Zhang W, Zhang LL, Luo ZP, Yang HL. Mid- to long-term results of total disc replacement for lumbar degenerative disc disease: a systematic review. J Orthop Surg Res. 2018 Dec 26;13(1):326. doi: 10.1186/s13018-018-1032-6. PMID 30585142
- [Background] Gornet MF, Burkus JK, Dryer RF, Peloza JH, Schranck FW, Copay AG. Lumbar disc arthroplasty versus anterior lumbar interbody fusion: 5-year outcomes for patients in the Maverick disc investigational device exemption study. J Neurosurg Spine. 2019 May 17;31(3):347-356. doi: 10.3171/2019.2.SPINE181037. Print 2019 Sep 1. PMID 31100723
- [Background] Panjabi M, Malcolmson G, Teng E, Tominaga Y, Henderson G, Serhan H. Hybrid testing of lumbar CHARITE discs versus fusions. Spine (Phila Pa 1976). 2007 Apr 20;32(9):959-66; discussion 967. doi: 10.1097/01.brs.0000260792.13893.88. PMID 17450069
- [Background] McAfee PC, Cunningham B, Holsapple G, Adams K, Blumenthal S, Guyer RD, Dmietriev A, Maxwell JH, Regan JJ, Isaza J. A prospective, randomized, multicenter Food and Drug Administration investigational device exemption study of lumbar total disc replacement with the CHARITE artificial disc versus lumbar fusion: part II: evaluation of radiographic outcomes and correlation of surgical technique accuracy with clinical outcomes. Spine (Phila Pa 1976). 2005 Jul 15;30(14):1576-83; discussion E388-90. doi: 10.1097/01.brs.0000170561.25636.1c. PMID 16025025
- [Background] Duan X, Shao Z, Xie K, Wang Z. [Research progress of percutaneous 360 degree axial lumbar interbody fusion technique]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2009 Aug;23(8):917-20. Chinese. PMID 19728605
- [Background] Li HM, Zhang RJ, Shen CL. Radiographic and Clinical Outcomes of Oblique Lateral Interbody Fusion Versus Minimally Invasive Transforaminal Lumbar Interbody Fusion for Degenerative Lumbar Disease. World Neurosurg. 2019 Feb;122:e627-e638. doi: 10.1016/j.wneu.2018.10.115. Epub 2018 Oct 26. PMID 31108079
- [Background] Ni J, Fang X, Zhong W, Liu N, Wood KB. Anterior Lumbar Interbody Fusion for Degenerative Discogenic Low Back Pain: Evaluation of L4-S1 Fusion. Medicine (Baltimore). 2015 Oct;94(43):e1851. doi: 10.1097/MD.0000000000001851. PMID 26512594
- [Background] Augusto A, Dias RG, Wajchenberg M, Martins D. EXTREME LATERAL INTERBODY FUSION IN PACIENTS WITH CHRONIC LOW BACK PAIN. Acta Ortop Bras. 2020 Sep-Oct;28(5):256-260. doi: 10.1590/1413-785220202805233621. PMID 33144843
- [Background] Hara M, Nishimura Y, Nakajima Y, Umebayashi D, Takemoto M, Yamamoto Y, Haimoto S. Transforaminal Lumbar Interbody Fusion for Lumbar Degenerative Disorders: Mini-open TLIF and Corrective TLIF. Neurol Med Chir (Tokyo). 2015;55(7):547-56. doi: 10.2176/nmc.oa.2014-0402. Epub 2015 Jun 29. PMID 26119895
- [Background] Lan T, Hu SY, Zhang YT, Zheng YC, Zhang R, Shen Z, Yang XJ. Comparison Between Posterior Lumbar Interbody Fusion and Transforaminal Lumbar Interbody Fusion for the Treatment of Lumbar Degenerative Diseases: A Systematic Review and Meta-Analysis. World Neurosurg. 2018 Apr;112:86-93. doi: 10.1016/j.wneu.2018.01.021. Epub 2018 Jan 31. PMID 29367001
- [Background] Parker LM, Murrell SE, Boden SD, Horton WC. The outcome of posterolateral fusion in highly selected patients with discogenic low back pain. Spine (Phila Pa 1976). 1996 Aug 15;21(16):1909-16; discussion 1916-7. doi: 10.1097/00007632-199608150-00016. PMID 8875725
- [Background] David T. Lumbar disc prosthesis. Surgical technique, indications and clinical results in 22 patients with a minimum of 12 months follow-up. Eur Spine J. 1993 Mar;1(4):254-9. doi: 10.1007/BF00298370. PMID 20054928
- [Background] Jacobs WC, van der Gaag NA, Kruyt MC, Tuschel A, de Kleuver M, Peul WC, Verbout AJ, Oner FC. Total disc replacement for chronic discogenic low back pain: a Cochrane review. Spine (Phila Pa 1976). 2013 Jan 1;38(1):24-36. doi: 10.1097/BRS.0b013e3182741b21. PMID 22996268
- [Background] Forsth P, Gerdhem P, Svensson O. [Lumbar disc prosthesis, a high risk treatment for low back pain.]. Lakartidningen. 2020 Mar 19;117:FZHI. Swedish. PMID 32242909
- [Background] Tobert DG, Antoci V, Patel SP, Saadat E, Bono CM. Adjacent Segment Disease in the Cervical and Lumbar Spine. Clin Spine Surg. 2017 Apr;30(3):94-101. doi: 10.1097/BSD.0000000000000442. PMID 27642820
- [Background] Bozduman O, Citir OC, Gurun E. Evaluation of Functional Capacity and Satisfaction of Patients With Lumbosacral Fusion. Cureus. 2023 Jan 27;15(1):e34284. doi: 10.7759/cureus.34284. eCollection 2023 Jan. PMID 36855476
- [Background] Drysch A, Ajiboye RM, Sharma A, Li J, Reza T, Harley D, Park DY, Pourtaheri S. Effectiveness of Reoperations for Adjacent Segment Disease Following Lumbar Spinal Fusion. Orthopedics. 2018 Mar 1;41(2):e161-e167. doi: 10.3928/01477447-20170621-02. Epub 2017 Jun 30. PMID 28662247
- [Background] Vraa ML, Myers CA, Young JL, Rhon DI. More Than 1 in 3 Patients With Chronic Low Back Pain Continue to Use Opioids Long-term After Spinal Fusion: A Systematic Review. Clin J Pain. 2021 Dec 1;38(3):222-230. doi: 10.1097/AJP.0000000000001006. PMID 34856579
- [Background] Koenders N, Rushton A, Verra ML, Willems PC, Hoogeboom TJ, Staal JB. Pain and disability after first-time spinal fusion for lumbar degenerative disorders: a systematic review and meta-analysis. Eur Spine J. 2019 Apr;28(4):696-709. doi: 10.1007/s00586-018-5680-3. Epub 2018 Jul 11. PMID 29995169
- [Background] Hashimoto K, Aizawa T, Kanno H, Itoi E. Adjacent segment degeneration after fusion spinal surgery-a systematic review. Int Orthop. 2019 Apr;43(4):987-993. doi: 10.1007/s00264-018-4241-z. Epub 2018 Nov 23. PMID 30470865
- [Background] Andersson GB, Mekhail NA, Block JE. Treatment of intractable discogenic low back pain. A systematic review of spinal fusion and intradiscal electrothermal therapy (IDET). Pain Physician. 2006 Jul;9(3):237-48. PMID 16886032
- [Background] Bydon M, De la Garza-Ramos R, Macki M, Baker A, Gokaslan AK, Bydon A. Lumbar fusion versus nonoperative management for treatment of discogenic low back pain: a systematic review and meta-analysis of randomized controlled trials. J Spinal Disord Tech. 2014 Jul;27(5):297-304. doi: 10.1097/BSD.0000000000000072. PMID 24346052
- [Background] DePalma MJ, Ketchum JM, Saullo TR, Laplante BL. Is the history of a surgical discectomy related to the source of chronic low back pain? Pain Physician. 2012 Jan-Feb;15(1):E53-8. PMID 22270748
- [Background] Zhao L, Manchikanti L, Kaye AD, Abd-Elsayed A. Treatment of Discogenic Low Back Pain: Current Treatment Strategies and Future Options-a Literature Review. Curr Pain Headache Rep. 2019 Nov 9;23(11):86. doi: 10.1007/s11916-019-0821-x. PMID 31707499
- [Background] Petersen T, Juhl CB, Fournier GL. Patients With Persistent Low Back Pain and Nerve Root Involvement: To Operate, or Not to Operate, That Is the Question. Spine (Phila Pa 1976). 2020 Apr 1;45(7):483-490. doi: 10.1097/BRS.0000000000003304. PMID 31658235
- [Background] Willems P. Decision making in surgical treatment of chronic low back pain: the performance of prognostic tests to select patients for lumbar spinal fusion. Acta Orthop Suppl. 2013 Feb;84(349):1-35. doi: 10.3109/17453674.2012.753565. PMID 23427903
- [Background] Mobbs RJ, Phan K, Malham G, Seex K, Rao PJ. Lumbar interbody fusion: techniques, indications and comparison of interbody fusion options including PLIF, TLIF, MI-TLIF, OLIF/ATP, LLIF and ALIF. J Spine Surg. 2015 Dec;1(1):2-18. doi: 10.3978/j.issn.2414-469X.2015.10.05. PMID 27683674
- [Background] Rahimzadeh P, Imani F, Ghahremani M, Faiz SHR. Comparison of percutaneous intradiscal ozone injection with laser disc decompression in discogenic low back pain. J Pain Res. 2018 Jul 31;11:1405-1410. doi: 10.2147/JPR.S164335. eCollection 2018. PMID 30104895
- [Background] Zeckser J, Wolff M, Tucker J, Goodwin J. Multipotent Mesenchymal Stem Cell Treatment for Discogenic Low Back Pain and Disc Degeneration. Stem Cells Int. 2016;2016:3908389. doi: 10.1155/2016/3908389. Epub 2016 Jan 11. PMID 26880958
- [Background] Mahmoudzadeh A, Rezaeian ZS, Karimi A, Dommerholt J. The effect of dry needling on the radiating pain in subjects with discogenic low-back pain: A randomized control trial. J Res Med Sci. 2016 Oct 18;21:86. doi: 10.4103/1735-1995.192502. eCollection 2016. PMID 28163732
- [Background] Manchikanti L, Pampati V, Kaye AD, Hirsch JA. Therapeutic lumbar facet joint nerve blocks in the treatment of chronic low back pain: cost utility analysis based on a randomized controlled trial. Korean J Pain. 2018 Jan;31(1):27-38. doi: 10.3344/kjp.2018.31.1.27. Epub 2018 Jan 2. PMID 29372023
- [Background] Helm Ii S, Simopoulos TT, Stojanovic M, Abdi S, El Terany MA. Effectiveness of Thermal Annular Procedures in Treating Discogenic Low Back Pain. Pain Physician. 2017 Sep;20(6):447-470. PMID 28934777
- [Background] Ko S, Vaccaro AR, Lee S, Lee J, Chang H. The prevalence of lumbar spine facet joint osteoarthritis and its association with low back pain in selected Korean populations. Clin Orthop Surg. 2014 Dec;6(4):385-91. doi: 10.4055/cios.2014.6.4.385. Epub 2014 Nov 10. PMID 25436061
- [Background] Simon J, McAuliffe M, Shamim F, Vuong N, Tahaei A. Discogenic low back pain. Phys Med Rehabil Clin N Am. 2014 May;25(2):305-17. doi: 10.1016/j.pmr.2014.01.006. Epub 2014 Feb 28. PMID 24787335
- [Background] Samini F, Gharedaghi M, Khajavi M, Samini M. The etiologies of low back pain in patients with lumbar disk herniation. Iran Red Crescent Med J. 2014 Oct 5;16(10):e15670. doi: 10.5812/ircmj.15670. eCollection 2014 Oct. PMID 25763198
- [Background] US Burden of Disease Collaborators; Mokdad AH, Ballestros K, Echko M, Glenn S, Olsen HE, Mullany E, Lee A, Khan AR, Ahmadi A, Ferrari AJ, Kasaeian A, Werdecker A, Carter A, Zipkin B, Sartorius B, Serdar B, Sykes BL, Troeger C, Fitzmaurice C, Rehm CD, Santomauro D, Kim D, Colombara D, Schwebel DC, Tsoi D, Kolte D, Nsoesie E, Nichols E, Oren E, Charlson FJ, Patton GC, Roth GA, Hosgood HD, Whiteford HA, Kyu H, Erskine HE, Huang H, Martopullo I, Singh JA, Nachega JB, Sanabria JR, Abbas K, Ong K, Tabb K, Krohn KJ, Cornaby L, Degenhardt L, Moses M, Farvid M, Griswold M, Criqui M, Bell M, Nguyen M, Wallin M, Mirarefin M, Qorbani M, Younis M, Fullman N, Liu P, Briant P, Gona P, Havmoller R, Leung R, Kimokoti R, Bazargan-Hejazi S, Hay SI, Yadgir S, Biryukov S, Vollset SE, Alam T, Frank T, Farid T, Miller T, Vos T, Barnighausen T, Gebrehiwot TT, Yano Y, Al-Aly Z, Mehari A, Handal A, Kandel A, Anderson B, Biroscak B, Mozaffarian D, Dorsey ER, Ding EL, Park EK, Wagner G, Hu G, Chen H, Sunshine JE, Khubchandani J, Leasher J, Leung J, Salomon J, Unutzer J, Cahill L, Cooper L, Horino M, Brauer M, Breitborde N, Hotez P, Topor-Madry R, Soneji S, Stranges S, James S, Amrock S, Jayaraman S, Patel T, Akinyemiju T, Skirbekk V, Kinfu Y, Bhutta Z, Jonas JB, Murray CJL. The State of US Health, 1990-2016: Burden of Diseases, Injuries, and Risk Factors Among US States. JAMA. 2018 Apr 10;319(14):1444-1472. doi: 10.1001/jama.2018.0158. PMID 29634829
- [Background] Becker BA, Childress MA. Nonspecific Low Back Pain and Return To Work. Am Fam Physician. 2019 Dec 1;100(11):697-703. PMID 31790184
- [Background] Luckhaupt SE, Dahlhamer JM, Gonzales GT, Lu ML, Groenewold M, Sweeney MH, Ward BW. Prevalence, Recognition of Work-Relatedness, and Effect on Work of Low Back Pain Among U.S. Workers. Ann Intern Med. 2019 Aug 20;171(4):301-304. doi: 10.7326/M18-3602. Epub 2019 May 14. PMID 31083729
- [Background] Yang H, Haldeman S, Lu ML, Baker D. Low Back Pain Prevalence and Related Workplace Psychosocial Risk Factors: A Study Using Data From the 2010 National Health Interview Survey. J Manipulative Physiol Ther. 2016 Sep;39(7):459-472. doi: 10.1016/j.jmpt.2016.07.004. Epub 2016 Aug 25. PMID 27568831
- [Background] Buchbinder R, van Tulder M, Oberg B, Costa LM, Woolf A, Schoene M, Croft P; Lancet Low Back Pain Series Working Group. Low back pain: a call for action. Lancet. 2018 Jun 9;391(10137):2384-2388. doi: 10.1016/S0140-6736(18)30488-4. Epub 2018 Mar 21. PMID 29573871
- [Background] Manchikanti L, Singh V, Falco FJ, Benyamin RM, Hirsch JA. Epidemiology of low back pain in adults. Neuromodulation. 2014 Oct;17 Suppl 2:3-10. doi: 10.1111/ner.12018. PMID 25395111
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Fatoye F, Gebrye T, Odeyemi I. Real-world incidence and prevalence of low back pain using routinely collected data. Rheumatol Int. 2019 Apr;39(4):619-626. doi: 10.1007/s00296-019-04273-0. Epub 2019 Mar 8. PMID 30848349